CLINICAL TRIAL: NCT02199873
Title: A Single Increasing Dose Safety, Tolerability and Pharmacodynamics (Methacholine Challenge) Study After Inhalational Administration of BIIX 1 XX (Single Doses: 5 - 800 mcg) in Healthy Young Male Volunteers (Randomised, Double-blind, Placebo-controlled)
Brief Title: Safety, Tolerability and Pharmacodynamics of BIIX 1 XX in Healthy Young Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1150.1
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BIIX 1 XX - single rising dose (Experimental)
  Interventions: Drug: BIIX 1 XX - single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIX 1 XX - single rising dose
  Arms: BIIX 1 XX - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety and tolerability of BIIX 1 XX, to determine the pharmacologically active dose (range) by performing a methacholine challenge test and to obtain preliminary pharmacokinetic data

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers who have Broca-Indices within +-20%
* Participants in the age range between 21 to 50 years
* Following the methacholine challenge the airway resistance (Raw) shows an increase of at least 130%
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteer is supposed to give his written informed consent prior to admission to the study
* As part of the screening (within 14 days before drug administration), each subject was to receive a complete medical examination (including blood pressure, pulse rate, medical history, documentation of demographics, inclusion/exclusion criteria and concomitant therapy) as well as a 12-lead Electrocardiogram (ECG)
* Haematopoietic, hepatic and renal function test will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration of the test substance

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (>= 24 hours) within one month before enrolment in the study
* Use of any drugs which might influence the results of the trial the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation within the last 4 weeks
* Excessive physical activities within the last week before the study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1998-06; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 3 months
Number of subjects with abnormal changes in laboratory parameters | up to 8 days after last drug administration
Change in impedance cardiography | up to 30 minutes after drug administration
Change in cutaneous microcirculation | up to 30 minutes after drug administration

SECONDARY OUTCOMES:
Change in airway resistance (Raw) after methacholine challenge | up to 30 minutes after drug administration
Change in specific conductance (sGaw) after methacholine challenge | up to 30 minutes after drug administration
AUC (Area under the concentration-time curve of the analyte in plasma) | up to 168 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 168 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 168 hours after drug administration
Ae (Amount of analyte that is eliminated in urine) | up to 48 hours after drug administration
MRT (Mean residence time of the analyte in the body) | up to 168 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 168 hours after drug administration
CL/F(Apparent clearance of the analyte in plasma following extravascular administration) | up to 168 hours after drug administration